CLINICAL TRIAL: NCT00679380
Title: Efficacy and Safety of Oral Budesonide-MMX™ (CB-01-02) 6 mg and 9 mg Extended Release Tablets in Patients With Mild or Moderate Active Ulcerative Colitis. A Multicentre, Randomised, Double-Blind, Double-Dummy, Comparative Study Versus Placebo With an Additional Reference Arm Evaluating Entocort®EC
Brief Title: (CB-01-02/02) Randomized Placebo Controlled Trial of Budesonide-multi-matrix System (MMX™) 6 mg and 9 mg in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Cosmo Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB-01-02/02
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Blood Specimen Collection; Endoscopy; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1: budesonide-MMX® 6 mg (Experimental): One budesonide-MMX® 6 mg plus three placebo Entocort EC® overencapsulated capsules daily in the morning after breakfast.
  Interventions: Procedure: Blood sampling, endoscopy; Drug: Budesonide MMX® 6 mg
- 2: budesonide-MMX® 9 mg (Experimental): One budesonide-MMX® 9 mg plus three placebo Entocort EC® overencapsulated capsules daily in the morning after breakfast.
  Interventions: Procedure: Blood sampling, endoscopy; Drug: Budesonide MMX® 9 mg
- 3: Entocort EC® 3 mg (Active Comparator): Three Entocort EC® 3 mg overencapsulated capsules plus one placebo budesonide MMX® tablet daily in the morning after breakfast.
  Interventions: Procedure: Blood sampling, endoscopy; Drug: Entocort EC® 3 mg
- 4: Placebo (Placebo Comparator): Three placebo Entocort EC® overencapsulated capsules plus one placebo Budesonide MMX® tablet daily in the morning after breakfast.
  Interventions: Procedure: Blood sampling, endoscopy; Drug: Placebo

INTERVENTIONS:
Procedure: Blood sampling, endoscopy — Blood sampling for hematology and biochemistry and endoscopy with biopsy for histological and endoscopic assessment scores
Drug: Budesonide MMX® 6 mg — 6 mg/day, 6 mg tablets
  Arms: 1: budesonide-MMX® 6 mg
Drug: Budesonide MMX® 9 mg — 9 mg/day, 9 mg tablets
  Arms: 2: budesonide-MMX® 9 mg
Drug: Entocort EC® 3 mg — 9 mg/day, 3 mg tablets
  Arms: 3: Entocort EC® 3 mg
Drug: Placebo — Placebo
  Arms: 4: Placebo

SUMMARY:
This will be a multicentre, randomised, double-blind, double-dummy, parallel group comparative study in patients with mild or moderate, active ulcerative colitis. The study will compare budesonide-MMX™ 6 mg and budesonide-MMX™ 9 mg tablets to placebo and to Entocort® 3 x 3 mg capsules, in four parallel groups of patients over an 8 week treatment period.

After the screening visit, patients will enter a washout period of 2 days, then they will be randomised to the following four treatment groups: budesonide-MMX™ tablets (6 mg), budesonide-MMX™ tablets (9 mg), Entocort® capsules (3 x 3 mg) and placebo (tablets and capsules), all administered once a day after breakfast. Hence, each patient will receive, in the morning after breakfast, either one budesonide-MMX™ 6 mg or budesonide MMX™ 9 mg tablet and 3 placebo Entocort® matching capsules, or three Entocort® 3 mg capsules and one placebo budesonide-MMX™ matching tablet, or one placebo budesonide-MMX™ matching tablet and three placebo Entocort® matching capsules.

DETAILED DESCRIPTION:
Each patient will receive one of the following regimens in the morning after breakfast:

1. One budesonide MMX® 6 mg tablet plus three placebo Entocort enteric-coated (EC®) overencapsulated capsules, or
2. One budesonide MMX® 9 mg tablet plus three placebo Entocort EC® overencapsulated capsules, or
3. Three placebo Entocort EC® overencapsulated capsules plus one placebo budesonide MMX® tablet, or
4. Three Entocort EC® 3 mg overencapsulated capsules plus one placebo budesonide MMX® tablet, daily for eight weeks.

Hence, each patient is to take four tablets/capsules per day of active or placebo study medication as per the randomization schedule. Placebo tablets of Budesonide MMX® and placebo overencapsulated capsules of Entocort EC® will be used to maintain the study blind using a double-dummy technique.

During the study, five visits to the clinical center are scheduled: one at Screening and three in the double-blind treatment period (Day 1, Day 14, Day 28 and Day 56). A safety follow-up visit will take place about 2 weeks after the final study visit. If a patient is withdrawn from the study before Day 56, they will be asked to attend the study center as soon as possible thereafter so that the Final visit assessments can be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the following criteria at the screening visit are eligible for participation in the study:

  * Male and female patients, 18-75 years old, suffering from ulcerative colitis for at least 6 months.
  * Diagnosis of ulcerative colitis in active phase, of mild or moderate entity with Ulcerative Colitis Disease Activity Index (UCDAI) ≥ 4 and ≤ 10 according to Sutherland.
  * All females of child-bearing potential must have a negative serum pregnancy test immediately prior to enrollment. In addition, all females of child-bearing potential must agree to be completely abstinent or be using an accepted form of contraception throughout the entire study period. Accepted forms of contraception are defined as those with a failure rate <1% when properly applied and include: combination oral pill, some intra-uterine devices, and a sterilised partner in a stable relationship. Female subjects must also not be actively breast-feeding through the entire study period.
  * Ability to comprehend the full nature and purpose of the study, including possible risks and side effects.
  * Ability to co-operate with the investigator and to comply with the requirements of the entire study.
  * Must be able to understand and voluntarily sign written informed consent prior to inclusion in the study.

Exclusion Criteria:

* Patients who meet any of the following criteria at screening visit are to be excluded from study participation:

  * Patients with limited distal proctitis (from anal verge up to 15 cm above the pectineal line).
  * Patients with severe ulcerative colitis (UCDAI >10).
  * Patients with infectious colitis.
  * Evidence or history of toxic megacolon.
  * Severe anaemia, leucopaenia or granulocytopaenia.
  * Use of oral or rectal steroids in the last 4 weeks.
  * Use of immuno-suppressive agents in the last 8 weeks before the study.
  * Use of anti tumour necrosis factor alpha (anti-TNFα) agents in the last 3 months.
  * Concomitant use of any rectal preparation.
  * Concomitant use of antibiotics.
  * Concurrent use of cytochrome P450 3A4 (CYP3A4) inducers or CYP3A4 inhibitors.
  * Patients with verified, presumed or expected pregnancy or ongoing lactation.
  * Patients with liver cirrhosis, or evident hepatic or renal disease or insufficiency, and/or severe impairment of the bio-humoural parameters (i.e. 2 x upper limit of normal for alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT) or creatinine).
  * Patient with severe diseases in other organs and systems.
  * Patients with local or systemic complications or other pathological states requiring a therapy with corticosteroids and/or immuno-suppressive agents.
  * Patients diagnosed with type 1 diabetes.
  * Patients diagnosed with, or with a family history of, glaucoma.
  * All patients with known hepatitis B, hepatitis C or with human immunodeficiency virus (HIV), according to the local privacy policy.
  * Participation in experimental therapeutic studies in the last 3 months. (Note: patients who participated in observational only studies are not excluded).
  * Any other medical condition that in the principal investigator's opinion would make the administration of the study drug or study procedures hazardous to the subject or obscure the interpretation of adverse events (AEs).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2008-06; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Travis, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (71):
- Australia (5):
  - Centre for Digestive Diseases, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide
  - Box Hill Hospital, Department of Gastroenterology Clive Ward Centre,, Box Hill
  - The Alfred Hospital, Melbourne
  - Monash Medical Centre, Melbourne
- Imelda Hospital, Bonheiden, Belgium
- Estonia (4):
  - East Viru Central Hospital, Kohtla-Järve
  - East Tallinn Central Hospital, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- France (2):
  - Hôpital Beaujon, Clichy
  - Hospital Saint-Louis, Paris
- Yaron Niv, Petah Tikva, Israel
- Italy (3):
  - CRO - IRCCS - Struttura Operativa Complessa di Gastroenterologia Oncologica, Aviano
  - Dipartimento di Medicina Interna e Specialità Mediche (DIMI), Genova
  - Divisione di Gastroenterologia - Istituto Clinico Humanitas IRCCS in Gastroenterologia, Milan
- Latvia (4):
  - Daugavpils Regional Hospital, Daugavpils
  - Paula Stradina Clinical University Hospital, Riga
  - Digestive Disease Centre Gastro, Riga
  - Clinical University Hospital Gailezers, Riga
- Lithuania (4):
  - Kaunas Medical University Hospital, Kaunas
  - Siauliai District Hospital, Šiauliai
  - M.Marcinkeviciaus Hospital, Vilnius
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Poland (13):
  - Niepubliczny Zaklad Opieki Zdrowotnej VIVAMED, Warsaw, Masovian Voivodeship
  - Centrum Leczenia Chorób Cywilizacyjnych, Warsaw, Masovian Voivodeship
  - Gastromed S.C., Bialystok, Podlaskie Voivodeship
  - Gastromed S.C.Maciej Kralisz, Andrzej Penpicki, Jacek Romatowski, Gabinet, Gastrologiczny i Pracownia Endoskopowa, Bialystok
  - NZOZ Centrum Leczenia Chorob Cywilizacyjnych, oddzial Gdynia, filia Fikakw, Gdynia
  - NZOZ Centrum Leczenia Chorob Cywilizacyjnych, Gdynia
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Szpital Uniwersytecki w Krakowie, Oddzial Kliniczny Kliniki Gastroenterologii, Hepatologii i Chorob Zakaznych,, Krakow
  - Szpital Uniwersytecki w Krakowie,Oddział Kliniczny Kliniki Gastroenterologii Hematologii i Chorób Zakaźnych, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej POLIMEDICA, Lodz
  - NZOZ Polimedica, Lodz
  - Endoskopia Sp. z o.o., Sopot
  - Endoskopia Sp.z o.o., Sopot
  - Indywidualna Specjalistyczna Praktyka Lekarska, Wejherowo
- Romania (4):
  - Spitalul Clinic Colentina Sectia Gastroenterologie, Bucharest
  - Cabinet Medical, Oradea
  - Spitalul Judetean Sibiu, Sibiu
  - Centrul de Gastroenterologie Dr. Goldis Adrian, Timișoara
- Russia (11):
  - Federal State Institution ?National Medical Surgical Center, Moscow
  - GU research educational medical centre of the administration of the affairs of the president of Russian Federation on the basis of State Healthcare Institution "State Clinical Hospital # 51", Moscow
  - State Scientific Centre of Coloproctology of the Federal Agency for High-Technology Medical Care, Moscow
  - GUZ of Moscow "City Clinical Hospital #24", Moscow
  - Rostov State Medical University, Rostov-on-Don
  - Saint-Petersburg GUZ City polyclinic #38 28, Saint Petersburg
  - Krestovsky Ireland Medical Institute, Saint Petersburg
  - FGU North-West DIstrict Medical Center of Roszdrav, Saint Petersburg
  - St. Petersburg State Medical Academy n.a. I.I. Mechnikov, Saint Petersburg
  - ZAO Clinic Dvizhenie, Volgograd
  - Yaroslavl Region Clinical Hospital, Yaroslavl
- Slovakia (4):
  - FNsP Bratislava, Nemocnica Stare Mesto 1st Internal Clinic Mickiewiczova, Bratislava
  - FNsP Bratislava, Nemocnica Ruzinov V. Interna klinika, Gastroenterohepatologicke oddelenie Ruzinovska, Bratislava
  - Gastroenterologické a Hepatologické centrum, Nitra
  - NsP Nove Mesto nad Vahom n.o., Nové Mesto nad Váhom
- Sweden (5):
  - Sahlgrenska Univerity Hospital, Gothenburg
  - Lund University Hospital, Lund
  - IBD-Unit, Sophiahemmet, Stockholm
  - Div. of Gastroenterology and Hepatology, Stockholm
  - Dept. of Gastroenerology and Hepatology, Stockholm
- Ukraine (6):
  - Chair of Gastroenterology and therapy of Dnipropetrovsk State Medical Academy based on Institute of gastroenterology, Dnipro
  - City Clinical Emergency Hospital named after O.I.Meschaninov,, Kharkiv
  - Lviv National Medical University after name Danylo Halytsky based on Communal Clinical City hospital No 5, Department of Propedeutic of Internal Disease, Lviv
  - Odessa city Polyclinic #20, Therapeutic Dept. 6, Odesa
  - Uzhgorod National University, Hospital surgery chair on the base of Uzhgorod Regional Clinical Hospital, Uzhhorod
  - Uzhgorod State Medical University, chair of therapy and family medicine, district clinical hospitalof station "Uzhgorod", Uzhhorod
- United Kingdom (4):
  - John Radcliffe Hospital, Headington, Oxford
  - University Hospital of Coventry and Warwickshire, Coventry
  - Gastrointestinal Unit, Edinburgh
  - St Marks Hospital, Harrow

REFERENCES:
- [Derived] Travis SP, Danese S, Kupcinskas L, Alexeeva O, D'Haens G, Gibson PR, Moro L, Jones R, Ballard ED, Masure J, Rossini M, Sandborn WJ. Once-daily budesonide MMX in active, mild-to-moderate ulcerative colitis: results from the randomised CORE II study. Gut. 2014 Mar;63(3):433-41. doi: 10.1136/gutjnl-2012-304258. Epub 2013 Feb 22. PMID 23436336

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from July 2008 to February 2010.
Pre-assignment Details: 3 randomized patients were not treated and are excluded from all analyses. The safety population, N= 511: 509 randomized and treated + 2 nonrandomized and treated patients. The intent-to-treat (ITT) population, N=410: 511 - 101 patients who were not randomized, had major entry criteria violation, GCP violation, or normal histology at baseline.
Period: Overall Study
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Entocort EC® 3 mg | 4: Placebo
Started | 109 | 109 | 103 | 89
Completed | 67 | 76 | 68 | 61
Not Completed | 42 | 33 | 35 | 28

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analyzed with the ITT population, defined as randomized patients who received study drug, had no entry criteria/GCP violation, and had abnormal mucosal histology at baseline. ITT population=410 patients: 511 - 101 patients who were not randomized, had entry criteria/GCP violation, or had normal histology at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Entocort EC® 3 mg | 4: Placebo | Total
Number analyzed (Participants) | 109 | 109 | 103 | 89 | 410
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 102 | 107 | 97 | 82 | 388
  >=65 years | 7 | 2 | 6 | 7 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (13.6) | 42.8 (13.9) | 43.4 (14.0) | 44.8 (13.0) | 43.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 45 | 48 | 32 | 177
  Male | 57 | 64 | 55 | 57 | 233
Region of Enrollment [Number; unit: participants]
  Estonia | 11 | 6 | 6 | 5 | 28
  Slovakia | 10 | 5 | 5 | 7 | 27
  Ukraine | 7 | 6 | 7 | 5 | 25
  Lithuania | 19 | 17 | 11 | 12 | 59
  Russian Federation | 24 | 35 | 34 | 28 | 121
  United Kingdom | 2 | 4 | 3 | 0 | 9
  Italy | 18 | 12 | 18 | 13 | 61
  France | 0 | 1 | 1 | 1 | 3
  Poland | 7 | 14 | 13 | 9 | 43
  Belgium | 2 | 0 | 0 | 0 | 2
  Romania | 2 | 5 | 1 | 3 | 11
  Australia | 1 | 1 | 3 | 2 | 7
  Latvia | 2 | 2 | 0 | 2 | 6
  Sweden | 3 | 1 | 0 | 2 | 6
  Israel | 1 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical and Endoscopic Remission.
Description: Clinical and endoscopic remission defined as an Ulcerative Colitis Disease Activity Index (UCDAI) score ≤ 1, with subscores of 0 for rectal bleeding, stool frequency, and mucosal appearance and with a ≥ 1 point reduction in the endoscopic index score.
Time Frame: 8 weeks
Population: Efficacy endpoints were analyzed with the ITT population, defined as randomized patients who received study drug, had no entry criteria/GCP violation, and had abnormal mucosal histology at baseline. ITT population=410 patients: 511 - 101 patients who were not randomized, had entry criteria/GCP violation, or had normal histology at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Entocort EC® 3 mg | 4: Placebo
Number analyzed (Participants) | 109 | 109 | 103 | 89
percentage of patients | 8.3 [3.1 to 13.4] | 17.4 [10.3 to 24.6] | 12.6 [6.2 to 19.0] | 4.5 [0.2 to 8.8]
Statistical Analysis 1: Comparison: 1: Budesonide-MMX® 6 mg vs 4: Placebo; All p-values were based on the Chi-square test; comparisons of budesonide MMX and placebo were conducted at the α = 0.025 level of significance and the comparison of Entocort EC and placebo were conducted at the α = 0.05 level of significance. The study was not powered to show statistical significance for Entocort EC versus budesonide MMX; Test type: Superiority or Other; p = 0.2876, Chi-squared; Difference in proportions = 3.8, 95% CI 2-sided [-3.0 to 10.5] — The difference in proportions was determined by subtracting the proportion of patients who reached the endpoint in the placebo group from that proportion in the active group (active minus placebo)
Statistical Analysis 2: Comparison: 2: Budesonide-MMX® 9 mg vs 4: Placebo; See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1); Test type: Superiority or Other; p = 0.0047, Chi-squared; Difference in proportions = 12.9, 95% CI 2-sided [4.6 to 21.3] — See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1)
Statistical Analysis 3: Comparison: 3: Entocort EC® 3 mg vs 4: Placebo; See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1); Test type: Superiority or Other; p = 0.0481, Chi-squared; Difference in proportions = 8.1, 95% CI 2-sided [0.4 to 15.9] — See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1)

2. Secondary Outcome: Clinical Improvement.
Description: Clinical improvement, defined as a ≥ 3-point improvement in UCDAI from baseline to the end of Week 8.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Entocort EC® 3 mg | 4: Placebo
Number analyzed (Participants) | 109 | 109 | 103 | 89
percentage of patients | 25.7 [17.5 to 33.9] | 42.2 [32.9 to 51.5] | 33.0 [23.9 to 42.1] | 33.7 [23.9 to 43.5]
Statistical Analysis 1: Comparison: 1: Budesonide-MMX® 6 mg vs 4: Placebo; Clinical improvement and endoscopic improvement were analyzed hierarchically. If at least one primary endpoint comparison was statistically significant, clinical improvement was to be compared between each budesonide MMX group and placebo at the α = 0.025 level of significance. If at least one comparison of clinical improvement was statistically significant, endoscopic improvement was to be compared between each budesonide MMX dose group and placebo at the α = 0.025 level of significance; Test type: Superiority or Other; p = 0.2174, Chi-squared; Difference in proportions = -8.0, 95% CI 2-sided [-20.8 to 4.] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 2: Budesonide-MMX® 9 mg vs 4: Placebo; See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1); Test type: Superiority or Other; p = 0.2215, Chi-squared; Difference in proportions = 8.5, 95% CI 2-sided [-5.0 to 22.0] — See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1)
Statistical Analysis 3: Comparison: 3: Entocort EC® 3 mg vs 4: Placebo; See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1); Test type: Superiority or Other; p = 0.9185, Chi-squared; Difference in proportions = -0.7, 95% CI 2-sided [-14.1 to 12.7] — See comments from the budesonide 6 mg versus placebo comparison (statistical analysis 1)

3. Secondary Outcome: Endoscopic Improvement.
Description: Greater or equal to a 1 point improvement in the mucosal appearance subscore of the UCDAI, from baseline to week 8.
  As per the hierarchical testing procedure for secondary endpoints, because clinical improvement was not statistically significant in the ITT population, formal statistical comparisons for endoscopic improvement between the 2 budesonide MMX groups and placebo were not conducted.
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Entocort EC® 3 mg | 4: Placebo
Number analyzed (Participants) | 109 | 109 | 103 | 89
percentage of patients | 25.7 [17.5 to 33.9] | 42.2 [32.9 to 51.5] | 36.9 [27.6 to 46.2] | 31.5 [21.8 to 41.1]
Statistical Analysis 1: Comparison: 3: Entocort EC® 3 mg vs 4: Placebo; As per the hierarchical testing procedure for secondary endpoints, because clinical improvement was not statistically significant in the ITT population, formal statistical comparisons for endoscopic improvement between the 2 budesonide MMX groups and placebo were not conducted. The statistical comparison between the Entocort EC and placebo groups is shown here; Test type: Superiority or Other; p = 0.4293, Chi-squared; Difference in proportions = 5.4, 95% CI 2-sided [-8.0 to 18.8] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 56 day ± 2 day (study duration) + 30 day safety followup period.
Description: Adverse event data were analyzed using the safety population, defined as all patients who received study drug. N= 511 for the safety population: 509 randomized and treated + 2 nonrandomized and treated patients.
Arm/Group | 1: Budesonide-MMX® 6 mg | 2: Budesonide-MMX® 9 mg | 3: Entocort EC® 3 mg | 4: Placebo
Serious Adverse Events (participants affected / at risk) | 3/128 | 4/128 | 1/126 | 5/129
Other Adverse Events (participants affected / at risk) | 77/128 | 67/128 | 68/126 | 52/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Budesonide-MMX® 6 mg (N=128) | 2: Budesonide-MMX® 9 mg (N=128) | 3: Entocort EC® 3 mg (N=126) | 4: Placebo (N=129)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Treatment failure (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Personality disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1: Budesonide-MMX® 6 mg (N=128) | 2: Budesonide-MMX® 9 mg (N=128) | 3: Entocort EC® 3 mg (N=126) | 4: Placebo (N=129)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (5) | 5 (6) | 7 (14) | 7 (7)
Abdominal pain upper (Gastrointestinal disorders) | 5 (9) | 3 (3) | 2 (2) | 3 (3)
Colitis ulcerative (Gastrointestinal disorders) | 20 (20) | 26 (26) | 15 (15) | 14 (14)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 4 (4) | 4 (7)
Flatulence (Gastrointestinal disorders) | 5 (7) | 7 (18) | 7 (16) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (10) | 6 (8) | 3 (7) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1) | 2 (2)
Treatment failure (General disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1) | 8 (9) | 6 (7) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Blood cortisol decreased (Investigations) | 7 (7) | 3 (3) | 4 (4) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Red blood cell sedimentation rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (3) | 4 (8) | 3 (7) | 1 (1)
Headache (Nervous system disorders) | 21 (30) | 20 (35) | 9 (15) | 8 (11)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3) | 4 (4) | 3 (4)
Mood altered (Psychiatric disorders) | 2 (2) | 0 (0) | 4 (4) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2) | 3 (3) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No